CLINICAL TRIAL: NCT02091752
Title: The ReTreatment Trial: A Phase II, Open-label, Single-arm Study of Re-treating Myelofibrosis Patients With Ruxolitinib/Jakavi After Treatment Interruption Due to Loss of Response and/or Adverse Event.
Brief Title: A Phase II Study of Re-treatment of Myelofibrosis Patients With Ruxolitinib/Jakavi After Treatment Interruption Due to Loss of Response and/or Adverse Event (ReTreatment Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to low enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2407
Record Dates: First submitted 2014-03-06; First posted 2014-03-19 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Primary Myelofibrosis
Keywords: Primary Myelofibrosis; Hematologic Diseases; Myeloproliferative Disorders; INC424; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis; Hematologic Diseases; Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): All participants received ruxolitinib.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Starting dose was based on reason for previous discontinuation of ruxolitinib (i.e. loss of response or AE) and baseline platelet count. For participants who previously discontinued ruxolitinib due to loss of response, the starting dose was determined based on baseline platelet counts as follows: participants with a baseline platelet count of ≥ 200 x 109/L began dosing at 20 mg po bid; participants with a baseline platelet count of 100 x 109/L to <200 x 109/L began dosing at 15 mg po bid. Participants who previously discontinued ruxolitinib due to an AE initiated therapy at a total daily dose 5 mg lower than the total daily dose prior to discontinuation.

SUMMARY:
The aim of the study is to assess the efficacy and safety of restarting ruxolitinib after treatment interruption due to loss of response and/or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PMF, PPV MF or PET-MF, irrespective of JAK2 mutational status according to the 2008 revised International Standard Criteria
* Peripheral blast count < 10%
* Requires therapy for MF in the opinion of the investigator
* Received prior monotherapy treatment with ruxolitinib for at least 12 consecutive weeks and experienced treatment interruption because of lossof response or adverse event
* Patients adhering to the Screening phase assessments and undergoing a a ruxolitinib-free washout period of a minimum of 1 week and a maximum of 8 weeks
* ECOG performance status 0, 1, 2, or 3
* Adequate bone marrow function
* Written informed consent

Exclusion Criteria:

* Patients not initially responding (primary resistance) to ruxolitinib therapy
* Patients who underwent a splenectomy or spleen radiation
* Patients currently scheduled for bone marrow transplant
* Patients who have discontinued ruxolitinib < 14 days prior to screening
* Patients who are not able to receive a starting dose of ruxolitinib of at least 15 mg total daily dose
* Leukemic transformation
* Inadequate renal function
* Presence of clinically meaningful active bacterial, fungal, parasitic or viral infection which requires therapy
* Previous history of Progressive Multifocal Leuko-encephalopathy (PML)
* Clinically significant cardiac disease or significant concurrent medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Leipzig, Germany
- Novartis Investigative Site, Florence, FI, Italy
- Novartis Investigative Site, Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated by Sponsor | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.00 (9.165)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving ≥20% Reduction From Baseline in Spleen Volume
Time Frame: Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Patients Achieving ≥35% Reduction From Baseline in Spleen Volume
Time Frame: Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Patients Achieving ≥25% and ≥50% Reduction, Respectively From Baseline, in Spleen Length
Time Frame: Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Spleen Length and Spleen Volume
Time Frame: Baseline, Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Patients Achieving ≥25% and ≥50% Reduction, Respectively, From Baseline in Total Symptom Score (MPN-SAF TSS)
Time Frame: Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in MPN-SAF TSS Score
Time Frame: Baseline, Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Time Frame: Week 1, Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and EuroQol (EQ)-5D-5L Scores
Time Frame: Baseline, Day 1, Week 8, Week 12, Week 16, Week 24
Population: The study was terminated early due to low enrollment. Analysis was not done.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ruxolitinib
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=3)
CONSTIPATION (Gastrointestinal disorders) | 1
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1
LISTERIOSIS (Infections and infestations) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1
CYSTITIS (Infections and infestations) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.